CLINICAL TRIAL: NCT01171807
Title: Dexamethasone Intra-Erythrocyte Therapy in Patients With Chron's Disease or Ulcerative Colitis
Brief Title: Erythrocytes-Mediated Delivery Of Dexamethasone 21-Phosphate In Steroid-Dependent Ulcerative Colitis
Acronym: Crocodex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quince Therapeutics S.p.A. (Industry)
Collaborators: Casa Sollievo della Sofferenza IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Crocodex; 2018-004763-31 (EudraCT Number)
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Steroid-dependency; Steroid adverse events; Erythrocytes
MeSH Terms: conditions — Colitis, Ulcerative | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Masking Description: No blinding procedures were applicable in this study which was designed as an open one.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dex 21-P (Experimental): In this arm a dose of 20 ml of Dex 2-P solution was administered every 15 or 30 days for a total of 3 or 6 treatment procedures, respectively.
  Specifically, steroid-dependant IBD patients had to undergo a total of 6 procedures at one month interval, while active mesalazine refractory UC patients had to undergo a total of 3 procedures at 15 days interval.
  Every procedure implies the collection and re-infusion of autologous erythrocytes previously loaded with Dex 21-P.
  Interventions: Drug: Dex 21-P
- Placebo (Placebo Comparator): In this arm placebo solution was administered every 15 or 30 days for a total of 3 or 6 treatment procedures, respectively.
  Specifically, steroid-dependant IBD patients had to undergo a total of 6 procedures at one month interval, while active mesalazine refractory UC patients had to undergo a total of 3 procedures at 15 days interval.
  Every procedure implies the collection and re-infusion of autologous erythrocytes previously NOT loaded with Dex21-P.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dex 21-P — At each procedure 50 ml of patient whole blood was washed with saline solution and centrifugated. The isolated erythrocytes were suspended into 2 hypotonic solutions to make their membrane permeable and incubated with Dex 21-P sodium salt up to obtain a final concentration of 10 mM. The drug loaded erythrocytes were immediately re-infused by using a suitable filter.
  Other Names: Dexamethasone 21-phosphate
  Arms: Dex 21-P
Drug: Placebo — Patients assigned to placebo arm performed the same procedure as the patients assigned to the DEX 21-P group without loading in the Red Blood Cells the Dex 21-P
  Arms: Placebo

SUMMARY:
Objectives:

The primary objective of this trial was to evaluate the patients response rate at the end of the study.

Patients were considered responder if one of the following conditions occurs:

* Disease remission (Powell Tuck ≤ 3 or CDAI < 150) and withdrawal of oral steroids therapy from at least the second treatment procedure;
* Disease marked improvement versus basal conditions (at least 5 point decrease in Powell Tuck index or 150 point decrease in CDAI score) and withdrawal of oral steroids therapy from at least the second treatment procedure.

Secondary objectives:

* to evaluate the endogenous cortisole production after receiving the study treatment
* to evaluate the inflammatory indexes (ESR and CPR) after receiving the study treatment
* to evaluate the endoscopic remission in patients suffering from mesalazine refractory Ulcerative Colitis
* to evaluate the safety of dexamethasone intra-erythrocyte therapy with particular attention to steroid-related adverse events.

DETAILED DESCRIPTION:
This was a single-center, placebo-controlled, randomised, phase II explorative study with the aim to investigate the ability of the new steroid delivery system to induce or maintain remission in steroid-dependent or mesalazine refractory patients suffering from Chron's disease (CD) or Ulcerative Colitis (UC) .

Once the patient was deemed eligible for the study, the treatment plan was selected as follows

In the Dexamethasone arm (DEX 21-P):

* steroid-dependant patients: one treatment procedure every 30 days up to a total of 6 procedures
* mesalazine refractory active UC patients: one treatment procedure every 15 days up to a total of 3 procedures.

In the placebo arm:

Patients assigned to placebo arm performed the same procedure as the patients assigned to the DEX 21-P group without loading in the Red Blood Cells the Dex 21-P.

The planned duration of individual patient participation in the study was a maximum of 6 or 28 weeks, depending from the assigned treatment scheme.

ELIGIBILITY:
Inclusion Criteria:

1. More than 18 years of age
2. Patients suffering from one of the following chronic inflammatory intestinal disease:

   * Steroid-dependent Chron's Disease or Ulcerative Colitis following ECCO definition or mild-moderate active UC ( Powell Tuck between 3 and 14- an index of 14 was allowed; endoscopic Baron score >1) refractory to mesalazine.
3. Disease extension over the rectum (at least 15 cm) in patients suffering from Ulcerative Colitis
4. Patients willing and be able to give written informed consent.

Exclusion Criteria:

1. Intestinal sub occlusion or a suspected abdomen abscess or a severe degree of the disease (CDAI > 450) in patient suffering from Chron's Disease
2. Patient affected by a severe Ulcerative Colitis (more than 6 evacuations of liquid, mucous-blooding stools combined at least one systemic sign as body temperature > 37.8 °C, heart rate < 90 bpm, ESR > 30 mm/h or haemoglobin < 10.5 g/dL)
3. Severe concurrent disease(s) as:

   * Medullar deficit: white blood cells < 3000/mm3; platelets < 75000/mm3; haemoglobin < 10 g/dL;
   * Hepatic diseases presenting total bilirubin ≥ 3 mg/dL; AST (GOT) ≥ 5 UNL; alkaline phosphatase ≥ 5 UNL:
   * Renal failure with serum creatinine ≥ 3 mg/dL;
   * Heart failure
   * Respiratory failure
   * Disabling neurological diseases
   * Neoplasia
   * Patient deemed candidate to surgery due to Chron's Disease or Ulcerative Colitis
   * Chronic alcohol or drug abuse
   * Patient for whom the use of steroids is contraindicated (e.g. systemic infections)
4. Treatment with Infliximab in the previous 4 months
5. Pregnant woman or female for whom the possibility of a pregnancy during the study could not be excluded.
6. Non-collaborating patient or subject unable to regularly undergo the scheduled study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-07-22 (Actual); Primary Completion 2007-05-15 (Actual); Study Completion 2007-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Andriulli, MD, Principal Investigator — Casa Sollievo della Sofferenza Hospital
Locations (1):
- Casa Sollievo della Sofferenza Hospital, San Giovanni Rotondo, Italy

REFERENCES:
- [Derived] Bossa F, Annese V, Valvano MR, Latiano A, Martino G, Rossi L, Magnani M, Palmieri O, Serafini S, Damonte G, De Santo E, Andriulli A. Erythrocytes-mediated delivery of dexamethasone 21-phosphate in steroid-dependent ulcerative colitis: a randomized, double-blind Sham-controlled study. Inflamm Bowel Dis. 2013 Aug;19(9):1872-9. doi: 10.1097/MIB.0b013e3182874065. PMID 23714676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total size of 40 patients was originally selected. However the final sample size of 33 was considered reasonable for the purpose of the study , due to the explorative nature of the protocol. Patients were assigned to a treatment plan consisting of a treatment procedure every 15 or 30 days for a total of 3 or 6 procedures, respectively.
Pre-assignment Details: Thirty-three (33) outpatients were enrolled into the study: nineteen subjects were steroid dependant (8 and 11 affected from Chron's Disease and Ulcerative Colitis, respectively) while 14 were patients with Ulcerative Colitis refractory to mesalazine.
Groups:
- Dex 21-P: In this arm a dose of 20 ml of Dex 2-P solution was administered every 15 or 30 days for a total of 3 or 6 treatment procedures, respectively.
  Specifically, steroid-dependant IBD patients had to undergo a total of 6 procedures at one month interval, while active mesalazine refractory UC patients had to undergo a total of 3 procedures at 15 days interval.
  Every procedure implies the collection and re-infusion of autologous erythrocytes previously loaded with Dex 21-P.
  Dex 21-P: At each procedure 50 ml of patient whole blood was washed with saline solution and centrifugated. The isolated erythrocytes were suspended into 2 hypotonic solutions to make their membrane permeable and incubated with Dex 21-P sodium salt up to obtain a final concentration of 10 mM. The drug loaded erythrocytes were immediately re-infused by using a suitable filter.
- Placebo: In this arm placebo solution was administered every 15 or 30 days for a total of 3 or 6 treatment procedures, respectively.
  Specifically, steroid-dependant IBD patients had to undergo a total of 6 procedures at one month interval, while active mesalazine refractory UC patients had to undergo a total of 3 procedures at 15 days interval.
  Every procedure implies the collection and re-infusion of autologous erythrocytes previously NOT loaded with Dex21-P.
  Placebo: Patients assigned to placebo arm performed the same procedure as the patients assigned to the DEX 21-P group without loading in the Red Blood Cells the Dex 21-P
Period: Overall Study
Arm/Group | Dex 21-P | Placebo
Started | 21 | 12
Intention to Treat (ITT) Population | 21 | 12
Per Protocol (PP) Population | 18 | 11
Safety (SAF) Population | 21 | 12
Completed | 15 | 8
Not Completed | 6 | 4
Not completed — Treatment failure | 2 | 4
Not completed — Non compliance | 1 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intention to Treat population (ITT): subjects who underwent at least one treatment procedure
Groups:
- Dex 21-P - ITT: In this arm a dose of 20 ml of Dex 2-P solution was administered every 15 or 30 days for a total of 3 or 6 treatment procedures, respectively.
  Specifically, steroid-dependant IBD patients had to undergo a total of 6 procedures at one month interval, while active mesalazine refractory UC patients had to undergo a total of 3 procedures at 15 days interval.
  Every procedure implies the collection and re-infusion of autologous erythrocytes previously loaded with Dex 21-P.
  Dex 21-P: At each procedure 50 ml of patient whole blood was washed with saline solution and centrifugated. The isolated erythrocytes were suspended into 2 hypotonic solutions to make their membrane permeable and incubated with Dex 21-P sodium salt up to obtain a final concentration of 10 mM. The drug loaded erythrocytes were immediately re-infused by using a suitable filter.
- Placebo - ITT: In this arm placebo solution was administered every 15 or 30 days for a total of 3 or 6 treatment procedures, respectively.
  Specifically, steroid-dependant IBD patients had to undergo a total of 6 procedures at one month interval, while active mesalazine refractory UC patients had to undergo a total of 3 procedures at 15 days interval.
  Every procedure implies the collection and re-infusion of autologous erythrocytes previously NOT loaded with Dex21-P.
  Placebo: Patients assigned to placebo arm performed the same procedure as the patients assigned to the DEX 21-P group without loading in the Red Blood Cells the Dex 21-P
- Total: Total of all reporting groups
Arm/Group | Dex 21-P - ITT | Placebo - ITT | Total
Number analyzed (Participants) | 21 | 12 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (10.1) | 40 (13.2) | 42 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 11 | 6 | 17
Region of Enrollment [Number; unit: participants]
  Italy | 21 | 12 | 33

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Responders to Dex 21-P vs Placebo
Description: Patients were considered responder if, at the EoS, one of the following occurred:
  * Disease remission (Powell Tuck index ≤ 3 or CDAI < 150) and withdrawal of oral steroids therapy from at least the second treatment procedure;
  * Disease marked improvement vs basal conditions (at least 5 point decrease in Powell Tuck or 150 point decrease in CDAI score) and withdrawal of oral steroids therapy from at least the second treatment procedure.
  The Powell-Tuck index was calculated by adding the subscores given by 7 items. A total score < 10 indicated a mild activity of the UC, and a total score >14 a severe one. The higher the score the worse the outcome.
  Crohn Disease Activity Index (CDAI) was a tool that combines subjective parameters, with objectives parameters. The score given to each parameter was inserted in an algorithm which provided the final Index value. A moderate CD showed a CDAI score between 220 and 450, while a CDAI > 450 was an activity index indicating a severe disease.
Time Frame: From baseline to End of treatment = 6 weeks ± 10 days (in chronic and steroid dependent IBD patients) or 28 weeks ± 5 days (in mesalazine refractory UC patients)
Population: ITT Population: subjects who underwent at least one treatment procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Dex 21-P - ITT | Placebo - ITT
Number analyzed (Participants) | 21 | 12
Participants
  Responders | 15 | 1
  Non Responders | 6 | 11
Statistical Analysis 1: Comparison: Dex 21-P - ITT vs Placebo - ITT; Test type: Superiority; p < 0.001, Chi-squared

2. Secondary Outcome: Change From Baseline in Endogenous Cortisole Blood Level After Receiving the Study Treatment
Description: Blood levels of endogenous cortisol were determined before the first and 15 days/one month after the last intra-erythrocytes infusion, according to the assigned treatment scheme planned for each patient. As steroids suppress ACTH production resulting in lowering cortisol levels, the assessment of this parameter was intended to investigate the ability of the dexamethasone intra-erythrocytes administration in minimising this steroid adverse effect.
  In child, from 1 to 16 years, the total serum cortisol reference range is 5-23 mcg/dL at 8 am, and 3-13 mcg/dL at 4 pm.
Time Frame: as for outcome 1
Population: Intent To Treat population (ITT): subjects who underwent at least one treatment procedure;
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Dex 21-P - ITT | Placebo - ITT
Number analyzed (Participants) | 21 | 12
mcg/dL | 3.3 (2.12) | 2.3 (5.71)

3. Secondary Outcome: Change From Baseline in Inflammatory Indexes After Receiving the Study Treatment: Erythrocyte Sedimentation Rate (ESR)
Description: The erythrocyte sedimentation rate (ESR) is the rate at which red blood cells in anticoagulated whole blood descend in a standardized tube over a period of one hour. It is a common hematology test, and is a non-specific measure of inflammation. To perform the test, anticoagulated blood is traditionally placed in an upright tube (Westergren tube) and the distance which the red blood cells fall is measured and reported in millimetres at the end of one hour. ESR was evaluated as supportive data for the assessment of the intestinal disease severity. It was determined before the first and 15 days/one month after the last intra-erythrocytes infusion, according to the assigned treatment scheme planned for each patient.
  ESR normal values in blood were from 0 to 20 mm/hour. Higher values are considered abnormal both in adults and in children. For ESR values > 100 mm/hour, there is a high probability that an underlying cause would be found upon investigation.
Time Frame: as for outcome 1
Population: Intent To Treat population (ITT): subjects who underwent at least one treatment procedure
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Dex 21-P - ITT | Placebo - ITT
Number analyzed (Participants) | 21 | 12
mm/h | -4.9 (25.88) | -9.3 (15.44)

4. Secondary Outcome: Change From Baseline in Inflammatory Indexes After Receiving the Study Treatment: C-reactive Protein (CRP)
Description: CRP is a protein produced by the liver. A C-reactive protein test measures the level of C-reactive protein (CRP) in a blood sample. Normal levels of blood C-reactive protein are low (0.3 to 1.0 mg/L). In case of inflammation liver releases more CRP into your bloodstream: results equal to or greater than 8 mg/L or 10 mg/L are considered high. High levels of CRP may indicate a serious health condition that causes inflammation.
  C-reactive protein (CRP) was determined before the first and 15 days/one month after the last intra-erythrocytes infusion, according to the assigned treatment scheme planned for each patient.
  Inflammation parameters (CRP) were evaluated as supportive data for the assessment of the intestinal disease severity.
  C-reactive protein was measured in milligrams per liter (mg/L). Results equal to or greater than 8 mg/L or 10 mg/L were considered high.
Time Frame: as for outcome 1
Population: Intent To Treat population (ITT): subjects who underwent at least one treatment procedure;
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Dex 21-P - ITT | Placebo - ITT
Number analyzed (Participants) | 21 | 12
mg/L | -0.5 (4.35) | -2.2 (7.27)

5. Secondary Outcome: Count of Partecipants, Suffering From Mesalazine Refractory UC, With Modification in Endoscopic Result (Baron Score)
Description: The Baron score was an endoscopic grading system for ulcerative colitis. Four grades are defined (0-3) by the Baron score according to the severity of macroscopic inflammation of the rectal mucosal appearances at rigid sigmoidoscopy: 0 = normal mucosa (ramifying vascular pattern clearly visible, no spontaneous bleeding, no bleeding to light touch);
  1. = abnormal mucosa but non-haemorrhagic appearances between scores 0 and 2;
  2. = moderately haemorrhagic (bleeding to light touch, but no spontaneous bleeding seen ahead of the instrument on initial inspection); 3= severely haemorrhagic (spontaneous bleeding seen ahead of instrument at initial inspection and bleeds to light touch).
  The higher the score the worst the outcome. Due to the nature of the score, its assessment was limited to patients suffering from UC, only. (CD or UC steroid-dependant patients were planned to receive the study treatment procedure every 30 days for a total of 6 administrations)
Time Frame: From baseline to End of treatment = 28 weeks ± 5 days (in mesalazine refractory UC patients)
Population: Intent To Treat population (ITT): subjects who underwent at least one treatment procedure.
  Herein only CD or UC steroid-dependant patients were analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dex 21-P - ITT | Placebo - ITT
Number analyzed (Participants) | 11 | 8
Participants
  From 0 to 0 score | 1 | 0
  From 1 to 0 score | 0 | 1
  From 1 to 1 score | 0 | 2
  From 1 to 2 score | 3 | 0
  From 2 to 1 score | 0 | 3
  From 2 to 2 score | 2 | 1
  From 3 to 1 score | 2 | 0
  From 3 to 2 score | 1 | 1
  From 3 to 3 score | 2 | 0

6. Secondary Outcome: Number of Patients Experiencing at Least One TEAE (Not Steroid-related)
Description: At each access to the clinic (except at the baseline visit one), patients were questioned and/or examined for evidence of adverse events. An adverse event was defined as any untoward medical occurrence or unfavourable and unintended sign in a subject administered a pharmaceutical product, biologic (at any dose), or medical device, whether or not considered related to the use of that product. This includes the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: as for outcome 1
Population: Safety Population: all patient included in ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Dex 21-P - SAF: In this arm a dose of 20 ml of Dex 2-P solution was administered every 15 or 30 days for a total of 3 or 6 treatment procedures, respectively.
  Specifically, steroid-dependant IBD patients had to undergo a total of 6 procedures at one month interval, while active mesalazine refractory UC patients had to undergo a total of 3 procedures at 15 days interval.
  Every procedure implies the collection and re-infusion of autologous erythrocytes previously loaded with Dex 21-P.
  Dex 21-P: At each procedure 50 ml of patient whole blood was washed with saline solution and centrifugated. The isolated erythrocytes were suspended into 2 hypotonic solutions to make their membrane permeable and incubated with Dex 21-P sodium salt up to obtain a final concentration of 10 mM. The drug loaded erythrocytes were immediately re-infused by using a suitable filter.
- Placebo - SAF: In this arm placebo solution was administered every 15 or 30 days for a total of 3 or 6 treatment procedures, respectively.
  Specifically, steroid-dependant IBD patients had to undergo a total of 6 procedures at one month interval, while active mesalazine refractory UC patients had to undergo a total of 3 procedures at 15 days interval.
  Every procedure implies the collection and re-infusion of autologous erythrocytes previously NOT loaded with Dex21-P.
  Placebo: Patients assigned to placebo arm performed the same procedure as the patients assigned to the DEX 21-P group without loading in the Red Blood Cells the Dex 21-P
Arm/Group | Dex 21-P - SAF | Placebo - SAF
Number analyzed (Participants) | 21 | 12
Participants
  Patients experiencing at least one TEAE | 11 | 8
  Patients experiencing at least one serious AE | 0 | 1

7. Secondary Outcome: Number of Patients Experiencing at Least One TEAE (Steroid-related)
Description: Steroid related adverse events were investigated to assess the ability of the therapeutic approach under study in reducing the occurrence or entity of steroid adverse effects.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dex 21-P - SAF | Placebo - SAF
Number analyzed (Participants) | 21 | 12
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: TEAEs were assessed throughout the study (except at the baseline visit 1) at each access to the clinic. More specifically adverse events were assessed: - steroid-dependant patients: every 30 days up to month 6 (Final Visit) - mesalazine refractory active UC patients: every 15 days up to 45 days (Final Visit)
Arm/Group | Dex 21-P - SAF | Placebo - SAF
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/12
Other Adverse Events (participants affected / at risk) | 11/21 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dex 21-P - SAF (N=21) | Placebo - SAF (N=12)
Acute pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dex 21-P - SAF (N=21) | Placebo - SAF (N=12)
Increase of alkaline phosphatase (Investigations) | 0 | 1
Increase on gamma-glutamyl transferase (Investigations) | 1 | 0
Increase of lipase (Investigations) | 2 | 0
Increase of amylase (Investigations) | 1 | 0
Joint aspiration (Investigations) | 0 | 1
Sideropenic anemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Loss of appetite (Metabolism and nutrition disorders) | 1 | 0
Weight decrease (Metabolism and nutrition disorders) | 1 | 0
Rectorrhage (Gastrointestinal disorders) | 0 | 2
Evacuations increase (Gastrointestinal disorders) | 0 | 2
Epigastralgia (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Tenesmus (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Rhinitis (Infections and infestations) | 1 | 0
Vertigo (Nervous system disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Hypotensive crisis (Injury, poisoning and procedural complications) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Articular pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Oedema (Vascular disorders) | 1 | 1
Shiver (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No